CLINICAL TRIAL: NCT01165671
Title: Randomized Phase II Study Evaluating a Carbon Ion Boost Applied After Combined Radiochemotherapy With Temozolomide Versus a Proton Boost After Radiochemotherapy With Temozolomide in Patients With Primary Glioblastoma
Brief Title: Carbon Ion Radiotherapy for Primary Glioblastoma
Acronym: CLEOPATRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEOPATRA; 2009-014668-21 (EudraCT Number); ISRCTN37428883 (Registry Identifier: BMC Study Registry)
Record Dates: First submitted 2010-07-13; First posted 2010-07-20 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2018-05

CONDITIONS: Primary Glioblastoma
Keywords: Primary Glioblastoma
MeSH Terms: interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): Carbon Ion Radiotherapy to the Macroscopic Tumor 6 x 3 Gy E up to 18 Gy E
  Interventions: Radiation: Carbon Ion Radiotherapy
- Standard Arm (Active Comparator): Proton Radiotherapy to the Macroscopic Tumor 5 x 2 Gy E up to 10 Gy E (Standard dose) applied after 48-52 Gy photon radiotherapy
  Interventions: Radiation: Proton Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Carbon ion Radiotherapy up to 18 Gy E in 3 Gy E fractions to the macroscopic tumor
  Arms: Experimental Arm
Radiation: Proton Radiotherapy — Proton Radiotherapy up to 10 Gy E in 2 Gy E fractions to the macroscopic tumor
  Arms: Standard Arm

SUMMARY:
Treatment standard for patients with primary glioblastoma (GBM) is combined radiochemotherapy with temozolomide (TMZ). Radiation is delivered up to a total dose of 60 Gy using photons. Using this treatment regimen, overall survival could be extended significantly however, median overall survival is still only about 15 months.

Carbon ions offer physical and biological advantages. Due to their inverted dose profile and the high local dose deposition within the Bragg peak precise dose application and sparing of normal tissue is possible. Moreover, in comparison to photons, carbon ions offer an increase relative biological effectiveness (RBE), which can be calculated between 2 and 5 depending on the GBM cell line as well as the endpoint analyzed. Protons, however, offer an RBE which is comparable to photons.

First Japanese Data on the evaluation of carbon ion radiation therapy showed promising results in a small and heterogeneous patient collective.

In the current Phase II-CLEOPATRA-Study a carbon ion boost will be compared to a proton boost applied to the macroscopic tumor after surgery at primary diagnosis in patients with GBM applied after standard radiochemotherapy with TMZ up to 50 Gy. In the experimental arm, a carbon ion boost will be applied to the macroscopic tumor up to a total dose of 18 Gy E in 6 fractions at a single dose of 3 Gy E. In the standard arm, a proton boost will be applied up to a total dose 10 Gy E in 5 single fractions of 2 Gy E.

Primary endpoint is overall survival, secondary objectives are progression-free survival, toxicity and safety.

DETAILED DESCRIPTION:
Study design

The purpose of the trial is to compare a carbon ion boost to a proton boost delivered to the macroscopic tumor in combination with combined radiochemotherapy with TMZ in patients with primary GBM.

The aim of the study is to compare overall survival as a primary endpoint, and progression free survival, toxicity and safety as secondary endpoints.

Focus of the analysis is to evaluate the change in overall survival and local control by carbon ion radiotherapy. Therefore, the aim of the trial is to evaluate the improvement in outcome due to effect of the altered biology of carbon ions on GBM. Chemotherapy with TMZ is considered standard treatment and is administered continuously as it would be applied in standard patient care outside any trial.

Trial Design The trial will be performed as a single-center two-armed randomized Phase II study.

Patients fulfilling the inclusion criteria will be randomized into two arms:

Arm A - Experimental Arm Carbon Ion Radiation Therapy as a Boost to the macroscopic tumor Total Dose 18 Gy E, 6 fractions, 3 Gy E single dose

Arm B - Standard Arm Proton Radiation Therapy as a Boost to the macroscopic tumor Total Dose 10 Gy E, 5 fractions, 2 Gy E single dose

Standard chemotherapy with TMZ will be continued during the experimental and standard arm in conventional dosing of 75 mg/m2 per day.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed unifocal, supratentorial primary glioblastoma
* macroscopic tumor after biopsy or subtotal resection
* indication for combined radiochemotherapy with temozolomide
* prior photon irradiation of 48-52 Gy to the T2-hyperintense area, resection cavity, areas of contrast enhancement adding 2-3cm safety margin in combination with standard temozolomide
* registration prior to photon RT or within photon RT allowing the beginning of particle therapy ≤ 4 days after completion of photon irradiation
* beginning of study treatment (proton or carbon ion RT) no later than 12 weeks after primary diagnosis
* age ≥ 18 years
* Karnofsky Performance Score ≥ 60
* adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the brain or chemotherapy with DTIC or TMZ other than during the radiochemotherapy stated in the inclusion criteria
* more than 52 Gy applied via photon-RT prior to particle therapy
* time interval of > 12 weeks after primary diagnosis (neurosurgical intervention) and beginning of study treatment (proton or carbon ion RT)
* Patients who have not yet recovered from acute toxicities of prior therapies
* Clinically active kidney, liver or cardiac disease
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 12 months

SECONDARY OUTCOMES:
Progression-free Survival | within 12 months
Toxicity | within 12 months
  CTCAC 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Department of Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Combs SE, Kieser M, Rieken S, Habermehl D, Jakel O, Haberer T, Nikoghosyan A, Haselmann R, Unterberg A, Wick W, Debus J. Randomized phase II study evaluating a carbon ion boost applied after combined radiochemotherapy with temozolomide versus a proton boost after radiochemotherapy with temozolomide in patients with primary glioblastoma: the CLEOPATRA trial. BMC Cancer. 2010 Sep 6;10:478. doi: 10.1186/1471-2407-10-478. PMID 20819220
- See also: Homepage Department of Radiation Oncology — http://www.klinikum.uni-heidelberg.de/ro